CLINICAL TRIAL: NCT01814033
Title: Use of the LRU Pillow in the Acute Setting Following Total Knee Arthroplasty
Acronym: LRU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newton-Wellesley Hospital (Other)
Responsible Party: Principal Investigator, Theresa J. Gustus, Rehabilitation Services Manager, Newton-Wellesley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRU1
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis
Keywords: LRU; Total Knee Arthroplasty; Total Knee Replacement; Acute Rehabilitation Total Knee; Total Knee Range of Motion; Total Knee Acute care Outcomes
MeSH Terms: conditions — Osteoarthritis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LRU Pillow (Experimental): Experimental: LRU Pillow
  Interventions: Other: Experimental: LRU Pillow
- Control Group (Active Comparator): Other: Control Group
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental: LRU Pillow — Foam wedge with a trough for positioning of the lower leg in an elevated position.
  Arms: LRU Pillow
Other: Control Group — Standard bed pillows placed under the lower leg to facilitate elevation
  Arms: Control Group

SUMMARY:
The Null Hypothesis is that there is no significant change in range of motion (ROM), pain, or function for a group of patients following total knee arthroplasty (TKA) who use the LRU pillow as compared to a control group of total knee arthroplasty patients who do not use the pillow.

DETAILED DESCRIPTION:
1. Study design will be a Pretest-Posttest Control Group Design . Enrollment would be random assignment of 20 patients to a control group vs 20 patients to a treatment group for patients with the diagnosis of osteoarthritis (OA) of the knee admitted for primary total knee arthroplasty. For specifics of patient assignment, please see below under Recruitment Procedures.
2. Unpaired t-Tests will be used to determine differences between mean scores for the dependent variables (pain, range of motion, functional mobility). Analysis of Covariance will be run to quantify the effect of the co-variates of age, gender, body mass index (BMI), and contralateral previous TKA. Confidence Intervals will be set at 95%.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee arthroplasty patients with primary diagnosis of osteoarthritis.

Exclusion criteria:

* bilateral total knee arthroplasties
* revision total knee arthroplasties
* unexpected decline in medical or mental status
* Subjects will range from 30 years of age to 80 years of age
* primary diagnosis of rheumatoid arthritis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 3 Days
  Knee ROM measured both actively and passively with a standard long arm goniometer twice daily for both groups.

SECONDARY OUTCOMES:
Pain | 3 Days
  Pain will be assessed using a visual analogue scale twice daily both at rest and with activity (exercise).

OTHER OUTCOMES:
Function | 3 Days
  Functional parameters of bed mobility, transfers, ambulation, gait, and stair climbing will be assessed daily using standard measures used in physical therapy assessment( dependent, moderate assist of one or two, minimal assist of one or two, hands on supervision, stand by supervision, or independence. )

CONTACTS AND LOCATIONS:
Overall Officials: Theresa J Gustus, PT, DPT, MS, Principal Investigator — Newton-Wellesley Hospital
Locations (1):
- Newton Wellesley Hospital, Newton, Massachusetts, United States

REFERENCES:
- [Background] Khanasuk Y, Ngarmukos S. Contemporary pain management in total knee arthroplasty. J Med Assoc Thai. 2012 Oct;95 Suppl 10:S238-44. PMID 23451469